CLINICAL TRIAL: NCT01532375
Title: Kochujang Decreases Visceral Fat and Improves Lipids Profiles
Brief Title: Kochujang, a Fermented Soybean-based Red Pepper Paste, Decreases Visceral Fat and Improves Blood Lipid Profiles in Overweight Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CUH_2008_AT_4
Record Dates: First submitted 2012-02-10; First posted 2012-02-14 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Overweight
Keywords: Kochujang,; visceral fat; population
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kochujang(32g) (Experimental)
  Interventions: Dietary Supplement: Kochujang
- placebo(32g) (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Kochujang — Kochujang (32g/day) for 12weeks.
  Arms: Kochujang(32g)
Dietary Supplement: placebo — placebo(32g/day) for 12weeks
  Arms: placebo(32g)

SUMMARY:
With the epidemic of obesity and diabetes growing around the world, Kochujang (KCJ) may be potentially effective in preventing and treating obesity and cardiovascular risks if proven in humans. However, human trial still have not been reported with KCJ supplementation. In the present study, we investigated the hypothesis that KCJ supplementation can be decrease the body fat and improve blood lipid profiles in overweight adults.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy of KCJ supplementation on anthropometric parameters, visceral fat/subcutaneous fat, and blood lipid profiles in overweight subjects.

Sixty overweight subjects with BMI >25 kg/m2 and waist-hip-ratio (WHR) ≥ 0.90 for men and ≥ 0.85 for women were randomly assigned to either KCJ supplement (n=30, 32 g/day) or placebo (n=30, 32 g/day) group for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI >25kg/m2 and 2)Waist-Hip Ratio (WHR): WHR> 0.90(male), WHR>0.85(female)

Exclusion Criteria:

* lipid metabolic disorders
* >10% changes in body weight in the past 3 months
* Cardiovascular disease such as arrhythmia, heart failure, myocardial infarction, and wearing pacemaker
* Allergy or hypersensitivity to any of the ingredients in the test products - History of reaction to any of the experimental products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* Participation in other clinical trials within the past 2 months
* Abnormal hepatic liver function, renal disease such as acute

  * chronic renal failure, nephrotic syndrome
* Use of anti-psychosis drug therapy within 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* History of alcohol or substance abuse
* Pregnancy or breastfeeding

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Visceral fat | after 12 weeks of consumption

SECONDARY OUTCOMES:
Body Mass Index | after 12 weeks of consumption
Subcutaneous fat | after 12weeks
Triglyceride | after 12week of consumption
Atherosclerosis index | after 12weeks of consumption
Apolipoprotein | after 12weeks of consumption

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Wan Chae, Ph.D, MD, Study Chair — Chonbuk National University Hospital

REFERENCES:
- [Derived] Cha YS, Kim SR, Yang JA, Back HI, Kim MG, Jung SJ, Song WO, Chae SW. Kochujang, fermented soybean-based red pepper paste, decreases visceral fat and improves blood lipid profiles in overweight adults. Nutr Metab (Lond). 2013 Feb 26;10(1):24. doi: 10.1186/1743-7075-10-24. PMID 23442518